CLINICAL TRIAL: NCT03866200
Title: Resveratrol Trial for Relief of Pain in Pseudoachondroplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit target number
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Karen Posey, Assoc. Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0573
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Pseudoachondroplasia
Keywords: resveratrol; joint pain
MeSH Terms: conditions — Pseudoachondroplasia; Arthralgia | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resveratrol, Then Placebo (Experimental): Participants first received Resveratrol 125 mg/day or 5 ml daily for 90 days. After a washout period of 30 days, they then received Placebo 5ml daily for 90 days.
  Interventions: Drug: resveratrol; Drug: Placebo
- Placebo, Then Resveratrol (Placebo Comparator): Participants first received Placebo 5ml daily for 90 days. After a washout period of 30 days, they then received Resveratrol 125 mg/day or 5 ml daily for 90 days.
  Interventions: Drug: resveratrol; Drug: Placebo

INTERVENTIONS:
Drug: resveratrol — 125 mg/day or 5 ml once per day for 90 days
  Other Names: resverages super berry tonic
Drug: Placebo — 5 ml once per day for 90 days

SUMMARY:
The purpose of this study is to determine if self-administered oral resveratrol can dampen joint pain for individuals with pseudoachondroplasia compared to placebo. Another goal of this study is to evaluate side effects in this population.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of pseudoachondroplasia is based on clinical assessment either in person or by photographic review by skeletal dysplasia specialist (JTH),
* Healthy beyond pseudoachondroplasia associated complications,

Exclusion Criteria:

* Current use of resveratrol
* Current use of blood thinners, lovastatin, ketoconazole, itraconazole, fexofenadine and triazolam.
* Other non-pseudoachondroplasia related health conditions, e.g. cancers.
* Pregnancy or breastfeeding. Women must use adequate contraception during the study.
* Participation in another clinical study and/or using investigational agents.
* Use of Non-steroid anti-inflammatory (NSAIDs) or aspirin.
* Current use of Alfentanil, Cyclosporine, Dihydroergotamine, Dofetilide, Ergotamine, Fentanyl, Flibanserin, Oxycodone, Pimavanserin, Pimozide, Quinidine, Saquinavir, Sirolimus, Tacrolimus, Temsirolimus, Theophylline, Tizanidine, Thioridazine, Fosphenytoin, Phenytoin or Warfarin.
* Baseline level of pain of 2 or higher on 10 point scale.
* Platelet count below 50,000 per ul on baseline complete blood count (CBC).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Posey, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Resveratrol, Then Placebo: Participants first received Resveratrol 125 mg/day or 5 ml daily for 90 days. After a washout period of 30 days, they then received Placebo 5ml daily for 90 days.
  resveratrol: 125 mg/day or 5 ml once per day for 90 days Placebo: 5 ml once per day for 90 days
- Placebo Comparator: Placebo, Then Resveratrol: Participants first received Placebo 5ml daily for 90 days. After a washout period of 30 days, they then received Resveratrol 125 mg/day or 5 ml daily for 90 days.
  resveratrol: 125 mg/day or 5 ml once per day for 90 days Placebo: 5 ml once per day for 90 days
Period: First Intervention (90 Days)
Arm/Group | Resveratrol, Then Placebo | Placebo Comparator: Placebo, Then Resveratrol
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0
Period: Washout (30 Days)
Arm/Group | Resveratrol, Then Placebo | Placebo Comparator: Placebo, Then Resveratrol
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0
Period: Second Intervention (90 Days)
Arm/Group | Resveratrol, Then Placebo | Placebo Comparator: Placebo, Then Resveratrol
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol, Then Placebo | Placebo, Then Resveratrol | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (16.36) | 49 (0) | 51.67 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain as Assessed by Numeric Pain Rating Scale
Description: total score 0-10 with higher scores indicating greater pain
Time Frame: baseline, 30 days, 60 days, 90 days
Population: Data were not collected for one participant
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Resveratrol: Participants who received Resveratrol 125 mg/day or 5 ml daily either the first or last 90 days of the study
- Placebo: Participants who received Placebo 5ml daily for either the first or last 90 days of the study.
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale
  Baseline | 3.60 (1.36) | 3.60 (1.36)
  30 days | 2.72 (1.24) | 2.36 (1.00)
  60 days | 2.44 (1.36) | 2.10 (1.09)
  90 days | 2.55 (0.92) | 1.92 (0.70)

2. Secondary Outcome: Health Related Quality of Life Score (HRQoL) Assessed by 36-item Short Form Health Survey Short Form-36 (SF-36)
Description: total score 0-100 with higher scores indicating better outcome
Time Frame: baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 68.60 (13.06) | 68.60 (13.06)
  30 days | 76.30 (11.23) | 75.84 (13.78)
  60 days | 70.17 (16.56) | 80.33 (13.46)
  90 days | 76.71 (14.27) | 77.54 (14.34)

ADVERSE EVENTS:
Time Frame: 90 days for each intervention
Arm/Group | Resveratrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03866200/Prot_SAP_000.pdf